CLINICAL TRIAL: NCT04826458
Title: Clinical Study Comparing Different Strategies to Increase Adherence to Oral Therapies in Oncohematology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRST100.28
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Solid Tumor; Hematologic Malignancy; Oral Drug Administration
Keywords: cancer; oral therapy; mobile app; electronic diary
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A. electronic diary (TreC-Onco) (Experimental): At the baseline visit, each patient assigned to arm A will be provided with the electronic diary (installed on a smart phone or tablet), the oral medication for the first treatment cycle and the appointment for the next cycle. The patient will be instructed on how to use the electronic diary, and the user manual will also be given. This app allows patients to record parameters related to their health state (e.g. medications, blood pressure, weight, fever, side effects or other symptoms) and through the "alarm" function, it reminds the patient to take the tablets, indicating the exact dosage. In addition, the patient can also indicate the dose reduction or the omission.
  Interventions: Device: TreC-Onco
- B. paper diary (Other): Patients assigned to arm B will be provided with a paper diary, oral medication for the first treatment cycle and the appointment for the next cycle. The patient will be instructed on how to use the paper diary.
  Interventions: Other: Paper diary

INTERVENTIONS:
Device: TreC-Onco — At the baseline visit, each patient assigned to arm A will be provided with the electronic diary (installed on a smart phone or tablet), the oral medication for the first treatment cycle and the appointment for the next cycle. The patient will be instructed on how to use the electronic diary, and the user manual will also be given. This app allows patients to record parameters related to their health state (e.g. medications, blood pressure, weight, fever, side effects or other symptoms) and through the "alarm" function, it reminds the patient to take the tablets, indicating the exact dosage. In addition, the patient can also indicate the dose reduction or the omission.
  Other Names: electronic diary
  Arms: A. electronic diary (TreC-Onco)
Other: Paper diary — Patients assigned to arm B will be provided with a paper diary, oral medication for the first treatment cycle and the appointment for the next cycle. The patient will be instructed on how to use the paper diary.
  Arms: B. paper diary

SUMMARY:
This is a multicenter, interventional, non-pharmacological study on a app for oral anticancer therapy management.

A total of 124 patients will be considered.

Patients will be randomized 1:1 to one of the following interventions:

A. electronic diary B. paper diary The primary aim of the study is to assess the effectiveness of the electronic diary in improving adherence to oral therapy treatment compared to the paper diary, in patients with solid and haematological tumors.

DETAILED DESCRIPTION:
This is a multicenter, interventional, non-pharmacological study on a app for oral anticancer therapy management.

The primary aim of the study is to assess the effectiveness of the electronic diary in improving adherence to oral therapy treatment compared to the paper diary, in patients with solid and haematological tumors.

The secondary objectives of the study are:

1. describe the reasons for non-adherence in each group (eg. forgetfulness, side effects, misunderstanding of prescription),
2. describe the patient's compliance with the instrument and modalities (electronic diary, paper diary) through a short questionnaire
3. description of the costs related to therapeutic non-adherence. A total of 124 patients will be considered: enrollment will take place consecutively until the predetermined number is reached.

Eligible patients will be randomized in a 1:1 ratio using a balanced procedure a blocks exchanged to one of the following interventions, stratified by type of therapy (chemotherapy vs. biological therapy): A. electronic diary B. paper diary The electronic diary consist of an Android app (for Android version 2.2 and later) for mobile devices, which acts as a diary for the patient.

Adherence will be assessed at each treatment cycle by counting the remaining tablets. For patients with disease progression within six treatment cycles, the assessment of adherence and therefore the count of the remaining tablets will end on the date of progression.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old (both genders)
* Eastern Cooperative Oncology Group (ECOG) ≤2
* Patients with solid and haematological neoplasia (adjuvant or advanced setting) candidates to treatment with oral therapy.

Exclusion Criteria:

* Patients who also receive anticancer treatment intravenously, as such patients access the hospital regularly and are in closer contact with healthcare personnel.
* Patients receiving experimental cancer treatment
* Patients who are unable to cooperate with study procedures (in the researcher's opinion)
* Patients who are candidates for oral drug treatment lasting less than 3 months.
* Patients with a life expectancy <12 weeks.
* All patients being treated with drugs not listed in the Protocol Appendix C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Adherence: drug accountability | 36 months
  To assess the effectiveness of the electronic diary in improving adherence to oral therapy.
  Adherence will be assessed at each treatment cycle by counting the remaining tablets, and tested using Fisher's exact test. The number of pills counted by the system will be compared with that counted by the physician as residual pills returned by the patient at the hospital visit.

SECONDARY OUTCOMES:
non-adherence reasons | 36 months
  to describe the reasons for non-adherence to treatment in each group (e.g. forgetfulness, side effects, misunderstanding of the prescription) through descriptive statistics: mean ± standard deviation (sd) or median and interquartile range for the variables continuous and absolute and relative frequency for categorical variables.
Patient compliance | 36 months
  describe the patient's compliance with the different strategies (paper diary or electronic) through a short questionnaire. Data are analysed through descriptive statistics: mean ± standard deviation (sd) or median and interquartile range for the variables continuous and absolute and relative frequency for categorical variables.
cost analysis | 36 months
  description of the costs associated with the lack of therapeutic adherence, both in terms of costs for drugs and overall health costs (hospitalizations, health services, access to the Emergency Department) (IRST center only). Data are analysed through descriptive statistics: mean ± standard deviation (sd) or median and interquartile range for the variables continuous and absolute and relative frequency for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Passardi, MD, Study Chair — IRCCS IRST
Locations (2):
- Italy (2):
  - Irst Irccs, Meldola, FC
  - Ospedale Civile Santa Chiara di Trento, Trento

IPD SHARING:
Plan to Share IPD: Yes
Data available for sharing: Individual participant data that underlie the results reported in the pubblication, after deindentification (text, tables, figures and appendices
Supporting Information: Study Protocol
Time Frame: Begining 9 months and ending 36 months following publication
Access Criteria: Proposals may be submitted up to 36 months after pubblication. URL will be provided on a later timepoint.

REFERENCES:
- [Derived] Passardi A, Serra P, Caffo O, Masini C, Brugugnoli E, Vespignani R, Giardino V, Petracci E, Bartolini G, Sullo F, Anesi C, Dianti M, Eccher C, Piras EM, Gios L, Campomori A, Oberosler V, Forti S. Use of the ONCO-TreC electronic diary compared with a standard paper diary to improve adherence to oral cancer therapy in patients with solid and haematological tumours: protocol for a randomised controlled trial. BMJ Open. 2022 Jan 11;12(1):e055814. doi: 10.1136/bmjopen-2021-055814. PMID 35017254